CLINICAL TRIAL: NCT01005953
Title: Phase 1 Study of a Digital/Internet/Mobile System for Collecting, Charting and Communicating About the Behaviors of Children on the Autism Spectrum
Brief Title: Comprehensive Collection, Charting, and Communication System
Acronym: CCCCSys
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: SymTrend Inc. (Industry)
Collaborators: University of Washington (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Minna Levine, PhD, SymTrend, Inc.
Other Study IDs: 1R41MH086153-01 (NIH)
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2011-06

CONDITIONS: Autism
Keywords: Autism; Behavioral Observations; Electronic diaries; Professionals treating children 3-10 with lower functioning autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Professionals treating autistic children: Special educators, occupational therapists, speech pathologists, behavior analysts who work with children on the spectrum.
- Families with autistic children (3-10)

SUMMARY:
As the prevalence of autism spectrum disorders continues to rise and the shortage of special education resources becomes more dramatic, the need for electronic tools that reduce the time burden of implementing an individual education plan (IEP) with pencil and paper methods becomes more apparent. SymTrend is going to expand its Internet and mobile computer/phone-based system for 1) collecting behavior data, 2) charting progress, 3) creating forms for #1 and #2, and 4) communicating within the IEP team, to include digital pen technology. Although this system will be tested with monitoring lower functioning children with autism, it has immediate relevance to a wide range of special education, mental health, and medical applications. The hypothesis is that this digital pen-based system will save time and money in the education of children on the spectrum and will enhance communication between schools and families.

DETAILED DESCRIPTION:
Project Summary: SymTrend is seeking funding to bring low-cost, technology-afforded power and efficiency to the special education (SPED) of a lower functioning child with autism (LFCA). Each LFCA has a federally mandated, individualized education plan (IEP). An effective IEP requires intensive school and home-based behavioral monitoring: iterations of behavioral data recording, progress charting, and team communication. SymTrend will extend the functionality of its current Internet and mobile system for behavioral monitoring to include the use of digital pen technology for recording on specially printed forms. The project will then test the two types of electronic monitoring (iPod Touch and digital pens) against current pencil and paper monitoring. It is hypothesized that an electronic system with four components - i.e., forms creation, data collection, progress charting, and team communication - will reduce the time burden of behavioral monitoring and enable schools to meet the IEP needs of its students within the constraints of very restrictive educational budgets.

Objectives: The three objectives of this project are 1) to design and implement a four-component behavioral monitor for IEPs that is easy-to-use, cost-sensitive, and has the power and efficiency to optimize and sustain behavioral improvement in LFCA; 2) to incorporate functionality for an extensive range of a) learning contexts, b) types of behavioral measurement, and c) progress charting formats that meet IEP reporting requirements; and 3) to contrast electronic behavioral monitoring with standard paper methods in terms of: a) efficiency, b) power, and c) acceptance.

Design and Methods: The test of the system will include a sample 15 children participating in one of two public school systems. LFCA will be monitored by parents and more than one type of professional both at school and at home. Monitoring will occur in the context of skill learning and disruptive behavior elimination. Professionals will keep track of their time and effort doing behavioral recording, charting, and communicating with other members of the IEP team. The research design includes within-subject comparisons of baseline paper monitoring versus electronic monitoring in terms of efficiency, power, and acceptance.

Significance: The electronic behavioral monitoring system created to support IEP use with LFCA can also be used with higher functioning children with autism (HFCA), other developmental disabilities (e.

g., ADHD), other clinical uses (e.g., depression and anxiety), academic use (e.g., university level behavioral science) and commercial use (e.g., human factors studies).

ELIGIBILITY:
Qualitative Professional Inclusion Criteria:

* Professional with licensure in one of the following professions (special education, occupational therapy, speech pathology, behavior analyst)
* Works professionally with children 3-10 with lower functioning autism in the home, in a clinic, or in a school
* Does behavioral observations and/or charting of treatment outcomes
* Able to get signed consent from parents of children seen by the professional, so that we can observe the professional.
* Has broadband Internet access.

Quantitative Professional Inclusion Criteria:

* Above criteria plus works in one of two schools conducting the research.

Exclusion Criteria:

* Have limited caseload in the two schools
* Work with children whose other professional colleagues working with those children are unwilling to participate (need at least two professionals/child)

Families - Qualitative Inclusion Criteria

* Have child 3-10 who has lower functioning autism (with appropriate documentation), who is seen by more than one professional.
* Has broadband Internet access

Families - Quantitative Inclusion Criteria

* Above criteria, plus has a child in one of the two programs participating in the study in Cambridge, MA and Newton, MA.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Qualitative Family Research: This research is open to families with children 3-10 with autism who have broadband Internet access at home or at work, whose children receive services from more than one caregiver (OT, special educator, speech pathologist, behavioral analyst/therapist).
  Qualitative Professional Research: This research is open to professionals working with children 3-10 with autism who have broadband Internet access and who keep detailed records about the work they do with their clients.
  Quantitative Research: Only open to families and professionals who are part of two school districts: Cambridge, MA and Newton, MA, who also meet the above criteria.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- SymTrend, Belmont, Massachusetts, United States

REFERENCES:
- See also: Description of SymTrend use with children with autism — https://www.symtrend.com/tw/public/public_docviewer?ltrans_doc=2166&no_title=true